CLINICAL TRIAL: NCT02601911
Title: Comparison of Ketorolac and Ketorolac/Acetaminophen on Success of Inferior Alveolar Nerve Block Injection
Brief Title: Effect of Premedication on Success of Inferior Alveolar Nerve Block Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nahid Mohammadzadeh Akhlaghi, Associate Professor, Azad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AzadUMS P/66/D
Record Dates: First submitted 2015-10-27; First posted 2015-11-11 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Irreversible Pulpitis
Keywords: Failure; Injection; Ketorolac; Premedication
MeSH Terms: interventions — Ketorolac Tromethamine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ketorolac tromethanine (Active Comparator): This group will receive a caplet including10 mg Ketorolac tromethamine 45 minutes before applying infra alveolar nerve block injection.
  Interventions: Drug: Ketorolac Tromethamine
- Acetaminophen (Active Comparator): This group receive a caplet including10 mg Ketorolac tromethamine/ 1000 mg Acetaminophen, before applying the injection.
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): This group receive a caplet including placebo, before applying the injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketorolac Tromethamine — 10 mg Ketorolac tromethamine is applied 45 minutes before the injection.
  Other Names: Toradol
  Arms: Ketorolac tromethanine
Drug: Acetaminophen — 10 mg Ketorolac tromethamine/ 1000mg Acetaminophen application before injection.
  Other Names: non
  Arms: Acetaminophen
Other: Placebo — This group receive the caplet including placebo 45 minutes before the injection.
  Arms: Placebo

SUMMARY:
The aim of this study is effect of premedication on success of inferior alveolar nerve block injection. Sixty healthy adult volunteers including criteria, are participating. The patients will be divided into 3 groups and will be randomly given one of premedications including 1) 10 mg Ketorolac, 2) 10 mg Ketorolac plus 1000mg Acetaminophen, and 3)Placebo, 45 minutes before applying the injection. All patients will receive standard Inferior Alveolar Nerve Block injection . Patients with no lip numbness and positive responses to cold and electric pulp tests would be excluded from the study. Endodontic access preparation will be initiated 15 minutes after Inferior Alveolar Nerve Block injection. Pain during treatment will be recorded using a Heft parker Visual Analog Scale(VAS). Success will be considered as no or mild pain (VAS≤54) during caries/dentin removal, access cavity preparation and working lengths measurements. Data will be analysed using Mann-U-Whitney and Kruskal-wallis tests.

DETAILED DESCRIPTION:
The aim of this study is effect of premedication on success of inferior alveolar nerve block injection. Sixty healthy adult volunteers with including criteria and with no spontaneous pain, reporting no or mild (Visual analog scale≤54) pain in response to cold testing and electric pulp tester, are participating. The patients will be divided into 3 groups on a random basis and will be randomly given one of the oral medications including 1) 10 mg Ketorolac, 2) 10 mg Ketorolac plus 1000mg Acetaminophen, and 3)Placebo, 45 minutes before applying the injection. All patients will receive standard Inferior Alveolar Nerve Block injection with one carpule of 4% Articaine with 1:100000 Epinephrine. Patients with no anesthetic sign (lip numbness) and positive responses to cold and electric pulp tests would be excluded from the study. Endodontic access preparation will be initiated 15 minutes after Inferior Alveolar Nerve Block injection. Pain during treatment will be recorded using a Heft parker Visual Analog Scale(VAS). Success will be considered as no or mild pain (VAS≤54) during caries/dentin removal, access cavity preparation and working lengths measurements. Data will be analysed using Mann-U-Whitney and Kruskal-wallis tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ranged 18-65
* without systemic diseases
* without any medicine consumption
* non smoking
* non pregnant
* non breast feeding
* with asymptomatic irreversible pulpitis ( Visual Analog Scale ≤ 54) in one mandibular molar that needs root canal treatment
* without any medicine consumption or analgesic and sedation
* understand and sign the VAS and consent forms

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain rate using Visual Analog Scale (VAS) form | 45 minutes
  Pain during caries and dentin removal , access cavity preparation and working lengths measurements using VAS form.

CONTACTS AND LOCATIONS:
Overall Officials: Nahid Mohammadzadeh Akhlaghi, DDS, MDS, Principal Investigator — Associate Professor
Locations (1):
- Dental Branch, AZad UMS, Tehran, Tehran Province, Iran